CLINICAL TRIAL: NCT06833528
Title: Assessment of the Clinical Performance of Novel Alkasite Restorative Material "Cention Forte" in Class II Restorations
Brief Title: Clinical Performance of Novel Alkasite Restorative Material "Cention Forte" in Class II Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ece Meral, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-23072
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries; Dental Caries Class II
Keywords: bioactive restorative materials; dental caries; alkasite
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cention Forte (Experimental): Self-etch primer will be applied. Cention Forte capsule will be activated, mixed, and directly applied. Light curing will be performed to accelerate polymerization.
  Interventions: Device: tooth restoration
- Composite Resin (Active Comparator): Selective enamel etching with 37% phosphoric acid for 15 seconds. G-Premio Universal Adhesive application. Incremental layering with light curing after each 2 mm layer.
  Interventions: Device: tooth restoration

INTERVENTIONS:
Device: tooth restoration — restoration of class II cavities
  Arms: Cention Forte
Device: tooth restoration — restoration of class II cavities
  Arms: Composite Resin

SUMMARY:
Background & Rationale:

Self-adhesive materials eliminate the need for adhesive protocols, offering advantages for direct restorations. The bulk-fill technique simplifies application by allowing a single-layer restoration. Glass ionomer cements (GICs) provide benefits such as fluoride release, remineralization, and moisture tolerance but have limitations, including poor aesthetics and low mechanical strength. To overcome these, hybrid materials combining GIC properties with composite durability have emerged.

Cention Forte, a capsulated alkasite restorative material, offers high flexural strength (>100 MPa), bioactivity, and ease of application. The manufacturer claims it is an ideal posterior restorative, potentially replacing composite resins and amalgam. Given that composite restorations fail more frequently in patients with isolation difficulties, limited mouth opening, or parafunctional habits, alternative materials are needed. This study evaluates Cention Forte as an alternative to conventional composites.

Objective:

To compare the clinical performance of Cention Forte with a universal composite resin (G-aenial Achord, GC) in Class II restorations over 18 months using FDI (World Dental Federation) criteria.

Hypothesis:

H₀: No significant difference between Cention Forte and composite resin after 18 months based on FDI criteria.

Primary Endpoint: At least 90% of restorations remain intact at 18 months with no significant differences in clinical performance.

Study Design:

A randomized, controlled, single-blind clinical trial with 30 healthy volunteers (18-35 years old), each receiving two restorations (one with Cention Forte, one with G-aenial Achord). Bite-wing radiographs will be taken before and after treatment, and at 6 , 12 and 18 months.

Eligibility Criteria:

Inclusion:

* 18-35 years old, systemically healthy.
* Brushing twice daily, at least 20 teeth in occlusion.
* At least two interproximal Class II lesions.
* Signed informed consent.

Exclusion:

* Pregnancy/lactation.
* Advanced periodontal disease, bruxism, malocclusion.
* Allergy to resin materials or local anesthesia.
* Endodontically treated teeth or pulp capping cases.

Restorative Procedure:

Study Group (Cention Forte):

Self-etch primer applied, followed by Cention Forte placement and light-curing.

Control Group (G-aenial Achord, GC):

Selective enamel etching with 37% phosphoric acid, followed by G-Premio Universal Adhesive and incremental layering with light-curing.

Clinical Evaluations (FDI Criteria):

Aesthetic properties: Color match, marginal discoloration, anatomical form. Functional properties: Fracture resistance, marginal adaptation, occlusal wear, proximal contact.

Biological properties: Postoperative sensitivity, secondary caries, periodontal response.

Scoring: 1 (excellent) to 5 (unacceptable).

Statistical Analysis:

Chi-square/Fisher's Exact Test: Compare clinical performance. Wilcoxon signed-rank test: Evaluate performance over time. Kaplan-Meier survival analysis: Assess restoration longevity. p < 0.05 considered statistically significant.

Ethical Considerations & Data Management:

Ethical approval from Hacettepe University Clinical Research Ethics Committee. Registration on ClinicalTrials.gov. Data secured and encrypted, accessible only to authorized personnel.

Expected Impact:

This study will assess whether Cention Forte is a viable alternative to composites, particularly for challenging clinical cases where isolation and durability are concerns.

DETAILED DESCRIPTION:
Background & Rationale The development of self-adhesive restorative materials has significantly improved clinical workflows by eliminating the need for separate adhesive protocols. In addition, the bulk-fill technique, which allows restorations to be completed in a single increment, provides a more efficient and user-friendly approach for posterior restorations.

Glass ionomer cements (GICs) have been widely used due to their fluoride release, remineralization capability, moisture tolerance, and cariostatic effects. However, they have notable limitations, such as inferior aesthetics, lower mechanical strength, and reduced wear resistance, which restrict their use as definitive restorative materials. Over the years, modifications have been made to improve GIC performance, including adding resins, altering the powder-to-liquid ratio, and incorporating metal reinforcements.

To address these limitations, hybrid restorative materials that combine the advantages of GICs (fluoride release, remineralization) with composite resin durability have been introduced. Among these materials is Cention Forte (Ivoclar), a capsulated alkasite restorative material designed for durability, ease of use, and bioactivity.

Cention Forte offers:

* High flexural strength (>100 MPa), exceeding the threshold for conventional posterior restorations.
* Remineralization properties, which prevent demineralization and enhance long-term restoration integrity.
* Aesthetic tooth-colored properties, overcoming the traditional drawback of GICs.
* Capsule formulation, improving handling compared to its predecessor, Cention N, which required manual mixing.

Given that composite resin restorations have lower success rates in patients with challenges such as isolation difficulties, limited mouth opening, or parafunctional habits, the Minamata Convention's restriction on dental amalgam use has further emphasized the need for an alternative restorative material. This study aims to compare the clinical performance of Cention Forte with a universal composite resin (G-aenial Achord, GC) in Class II restorations over a 12-month follow-up period.

Study Objective The primary objective is to evaluate and compare the clinical performance of Cention Forte and G-aenial Achord (GC) in Class II posterior restorations using the FDI World Dental Federation criteria over 12 months.

Study Hypothesis Null Hypothesis (H₀): There will be no significant difference between Cention Forte and the universal composite resin based on FDI criteria at the end of 18 months.

Primary Endpoint: At least 90% of restorations remain intact after 18 months, with no significant differences in clinical performance.

Study Design This study is designed as a randomized, controlled, single-blind clinical trial. Participants will undergo a split-mouth design, where each individual receives two restorations: one with Cention Forte and the other with G-aenial Achord.

Study Center: Hacettepe University Faculty of Dentistry Study Duration: 18 months Sample Size: 38 volunteers (18-35 years old), each receiving two Class II restorations (total: 76 restorations) Randomization: The Research Randomizer Program will be used to allocate teeth into three restorative groups.

Eligibility Criteria

Inclusion Criteria:

* Healthy individuals aged 18-35 years
* Brushing twice daily and maintaining good oral hygiene
* At least two interproximal Class II carious lesions in molar teeth
* At least 20 teeth in occlusion with antagonist contacts
* Signed informed consent and completion of initial periodontal therapy

Exclusion Criteria:

* Pregnancy or lactation
* Advanced periodontal disease
* Bruxism or malocclusion
* Allergy to resin-based materials or local anesthesia
* Endodontically treated teeth or those requiring pulp capping

Restorative Procedures

1. Cavity Preparation

   Standardized Class II cavities will be prepared with dimensions ensuring the lesions remain within enamel and dentin.

   Bite-wing radiographs will be taken before treatment to assess lesion depth and proximity to the pulp.

   Rubber dam or cotton roll isolation will be used to control moisture.
2. Study Group (Cention Forte):

   Self-etch primer will be applied. Cention Forte capsule will be activated, mixed, and directly applied. Light curing will be performed to accelerate polymerization.
3. Control Group (G-aenial Achord, GC):

Selective enamel etching with 37% phosphoric acid for 15 seconds. G-Premio Universal Adhesive application. Incremental layering with light curing after each 2 mm layer. Clinical Evaluations

Restorations will be assessed immediately after placement, at 6 months, and at 18 months using the FDI criteria, which include:

1. Aesthetic Properties:

   Color match and stability Marginal discoloration Anatomical form
2. Functional Properties:

   Fracture resistance Marginal adaptation Occlusal wear Proximal contact integrity
3. Biological Properties:

Postoperative sensitivity Secondary caries development Periodontal response Restorations will be photographed and scored from 1 (excellent) to 5 (unacceptable).

Statistical Analysis Chi-square or Fisher's Exact Test: Compare clinical performance of both materials.

Wilcoxon Signed-Rank Test: Evaluate time-based changes in FDI scores. Kaplan-Meier Survival Analysis: Assess restoration longevity. p < 0.05 will indicate statistical significance. Ethical Considerations & Data Management Ethical approval from the Clinical Research Ethics Committee of Hacettepe University.

Study registration on ClinicalTrials.gov to ensure transparency and compliance with ethical guidelines.

Patient data and photographs will be securely stored in an encrypted system, accessible only to authorized personnel.

Expected Impact This study aims to determine whether Cention Forte can serve as a viable alternative to composite resins for posterior Class II restorations, particularly in challenging clinical scenarios. If successful, Cention Forte could provide a more durable, bioactive, and easy-to-use restorative option, reducing failures in cases with limited isolation or high caries risk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-35 years

  * Brushing twice daily and maintaining good oral hygiene
  * At least two interproximal Class II carious lesions in molar teeth
  * At least 20 teeth in occlusion with antagonist contacts
  * Signed informed consent and completion of initial periodontal therapy

Exclusion Criteria:

* Pregnancy or lactation

  * Advanced periodontal disease
  * Bruxism or malocclusion
  * Allergy to resin-based materials or local anesthesia
  * Endodontically treated teeth or those requiring pulp capping

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Retention Alpha for at least 90% of the restorations | 18 months
  The primary factor for determining the clinical performance of a restorative material is the retention rate. It represents the survival rates of the restorations after a period of time. According to ADA guidelines, a restorative material should show at leat 90% alpha retention rate after 18 months to be considered as clinically acceptable. The retention is assesed as alpha (retentive restoratation) or charlie (failed restoration). Clinical evaluation is performed to examine if the restoration is in place or has fallen.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided